CLINICAL TRIAL: NCT03345745
Title: The Short-Term Effects of Non-Surgical Periodontal Therapy on The Saliva Levels of S100A12, High-Sensitivity C-Reactive Protein and Fetuin-A in Patients With Gingivitis and Chronic Periodontitis
Brief Title: Saliva Levels of S100A12, CRP, Fetuin-A in Periodontal Disease Patients
Status: Completed | Type: Observational
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Cankat Kara, Professor, Ordu University
Other Study IDs: OrduUniversityDentistry
Record Dates: First submitted 2017-11-13; First posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Periodontal Inflammation
Keywords: Fetuin-A; S100A12; C-Reactive Protein; Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Periodontally healthy subjects: Salivary samples
  Interventions: Diagnostic Test: salivary samples
- Chronic periodontitis patients: Salivary samples
  Interventions: Diagnostic Test: salivary samples
- Gingivitis patients: Salivary samples
  Interventions: Diagnostic Test: salivary samples

INTERVENTIONS:
Diagnostic Test: salivary samples — Salivary Hs-CRP, Fetuin-A and S100A12 levels and salivary flow rates were evaluated at baseline and a month after the treatments

SUMMARY:
Hs-CRP, Fetuin-A and S100A12 are acute phase proteins associated with many systemic diseases and conditions. The aim of this study was to determine the clinical parameters and salivary Hs-CRP, Fetuin-A and S100A12 levels before and after non-surgical periodontal treatments in the patients with periodontal diseases.

A total of 54 subjects were divided in to three groups; periodontally healthy (n: 18), gingivitis (n: 18), chronic periodontitis (n: 18). Clinical periodontal parameters, salivary Hs-CRP, Fetuin-A and S100A12 levels and salivary flow rates were evaluated at baseline and a month after the treatments. Salivary Hs-CRP, Fetuin-A and S100A12 levels were assayed by ELISA.

ELIGIBILITY:
Inclusion Criteria:

never-smokers no history of systemic disease no patients had been under periodontal therapy and medicine for at least 6 months before the study no pregnancy or lactation no alcohol or antioxidant vitamin consumption.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Fifty-four patients (27 women) aged 25-45 years who had presented to our faculty for periodontal and other dental problems and consented to participate were enrolled in the study.
  Group 1 - subjects with healthy periodontal status Group 2 - subjects with untreated gingivitis Group 3 - subjects with untreated chronic periodontitis (indicted by radiographic evidence of bone loss and clinical attachment loss > 5 mm in more than six teeth)
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Salivary acute phase proteins | Baseline - a month after the periodontal treatments
  Fetuin-A
Salivary acute phase proteins | Baseline - a month after the periodontal treatments
  S100A12
Salivary acute phase proteins | Baseline
  C-Reactive Protein

SECONDARY OUTCOMES:
Evaluating periodontal health | Baseline - a month after the periodontal treatments
  plaque index
Evaluating periodontal health | Baseline - a month after the periodontal treatments
  gingival index
Evaluating periodontal health | Baseline
  probing depth
Evaluating periodontal health | Baseline - a month after the periodontal treatments
  clinical attachment level
Evaluating periodontal health | Baseline - a month after the periodontal treatments
  gingival bleeding on probing

CONTACTS AND LOCATIONS:
Locations (1):
- Ordu University, Ordu, Turkey (Türkiye)